CLINICAL TRIAL: NCT04926844
Title: Effectiveness of Combined Levetiracetam and Midazolam in Treatment of Generalized Convulsive Status Epilepticus in Children
Brief Title: Effectiveness of Combined Levetiracetam and Midazolam in Generalized Convulsive Status Epilepticus in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelhamid Elshater, Pediatric Resident, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Soh-Med-21-06-07
Record Dates: First submitted 2021-06-14; First posted 2021-06-15 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Status Epilepticus; Generalized Convulsive Status Epilepticus; Status Epilepticus, Generalized; Status Epilepticus, Generalized Convulsive
Keywords: Status epilepticus; Convulsions; Children; Seizures; Benzodiazepines; Midazolam; Levetiracetam
MeSH Terms: conditions — Status Epilepticus; Seizures | interventions — Levetiracetam; Midazolam

STUDY DESIGN:
Intervention Model Description: Two groups of children with continuing seizures after stabilization phase (5 minutes):
  1. Study group; will receive intravenous levetiracetam 60 mg/kg (max 4500 mg) over 5 minutes (diluted with isotonic saline to a concentration of 50 mg/ml).
  2. Control group will receive intravenous isotonic saline (as a placebo) in the same way. At the same time, both groups will receive intravenous midazolam 0.2 mg/kg (maximum 10 mg) over 2 minutes.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each enrolled child will be assigned a unique identification number. Pharmacy will fill the active and placebo preparations in similar containers with sealed code for identification. Participants' families, treating clinicians, and investigators will be unaware of group assignment and drug/placebo therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Children receiving levetiracetam + midazolam
  Interventions: Drug: Levetiracetam; Drug: Midazolam
- Control group (Placebo Comparator): Children receiving placebo + midazolam
  Interventions: Drug: Midazolam; Drug: Placebo

INTERVENTIONS:
Drug: Levetiracetam — Intravenous levetiracetam 60 mg/kg (max 4500 mg) over 5 minutes (diluted with isotonic saline to a concentration of 50 mg/ml).
  Other Names: Keppra; Tiratam
  Arms: Study group
Drug: Midazolam — Intravenous midazolam 0.2 mg/kg (maximum 10 mg) over 2 minutes
Drug: Placebo — Intravenous isotonic saline (1.2 ml/kg) over 5 minutes
  Arms: Control group

SUMMARY:
Generalized status epilepticus is a common pediatric neurological emergency with significant mortality and morbidity. Benzodiazepines remain the first anticonvulsive line but benzo-diazepines don't control seizures in about 30% of cases. GCSE may be more rapidly stopped and controlled through combining another drug with benzodiazepines such as Levetiracetam, acting by different pathways. This study aims to evaluate the effectiveness of combined levetiracetam and midazolam in treatment of generalized convulsive status epilepticus in children.

DETAILED DESCRIPTION:
Generalized convulsive status epilepticus (GCSE) is a common pediatric neurological emergency with an annual incidence of up to 73 episodes per 100,000 children and is associated with mortality in 2.7% of cases and overall morbidity in 10% - 20% of cases, including hemodynamic instability and long-term neurological impairments.

The management of GCSE in children starts with emergency measures (stabilization phase) with monitoring and laboratory testing in the first 5 minutes. Benzodiazepines are used as first-line anticonvulsants for GCSE that persists for more than 5 minutes. However, studies have shown that benzo-diazepines don't control GCSE in about 30% of patients. GCSE may be more rapidly stopped and controlled through combining another drug with benzodiazepines, acting by different pathways.

Levetiracetam is a recent broad-spectrum antiepileptic drug with a relatively high safety profile. The effectiveness of intravenous levetiracetam has been demonstrated as a second-line anticonvulsant in GCSE. In this study, we aim to evaluate the effectiveness and safety of levetiracetam plus midazolam versus midazolam alone as first-line therapy of GCSE in children.

ELIGIBILITY:
Inclusion Criteria:

* Generalized convulsive status epilepticus, which is clinically defined at the time of presentation as continuous, generalized, tonic-clonic seizure activity or ≥ 2 generalized tonic-clonic seizures without recovery of consciousness for more than 5 minutes.

Exclusion Criteria:

* Failure to obtain informed consent.
* Prior therapy with any anticonvulsant for the presenting episode of generalized convulsive status epilepticus.
* Epileptic patients on levetiracetam therapy.
* Known allergy or contraindications to any of the study drugs.
* End-stage kidney disease.
* Severe liver disease.
* Cardiac diseases.
* Hypoglycemia or hyperglycemia.
* Inborn errors of metabolism.
* Known mood/behavioral disorder.
* Failure to obtain intravenous access in the first 5 minutes.
* Cessation of seizures during the stabilization phase (0 - 5 minutes).
* Traumatic brain injury

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2021-06-20 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Cessation of seizures | 20 minutes
  Cessation of clinical seizures at 20 minutes timepoint (end of first therapy phase)

SECONDARY OUTCOMES:
Need for repeating midazolam | 20 minutes
  Need for repeating midazolam during the first therapy phase (5 - 20 min)
Cessation of seizures | 40 minutes
  Cessation of clinical seizures at 40 minutes timepoint (end of second therapy phase).
Seizure control | 24 hours
  24-hours seizure control (no visually observed recurrence of seizures after the end of second phase therapy with improved sensorium)
Hypotension | 24 hours
  Occurrence of hypotension
Need for mechanical ventilation | 24 hours
  Need for mechanical ventilation
Skin rash | 24 hours
  Occurrence of skin rash
Agitation/aggression | 24 hours
  Occurrence of agitation/aggression
Mortality | 24 hours
  Occurrence of death

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrahim A Sadek, MD, PhD, Study Chair — Sohag University
Locations (1):
- Department of Pediatrics - Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Unidentified individual patients' data will be available on resonable request after publication
Supporting Information: Study Protocol
Time Frame: After publication for 3 years
Access Criteria: Contact the principal investigator

REFERENCES:
- [Background] Glauser T, Shinnar S, Gloss D, Alldredge B, Arya R, Bainbridge J, Bare M, Bleck T, Dodson WE, Garrity L, Jagoda A, Lowenstein D, Pellock J, Riviello J, Sloan E, Treiman DM. Evidence-Based Guideline: Treatment of Convulsive Status Epilepticus in Children and Adults: Report of the Guideline Committee of the American Epilepsy Society. Epilepsy Curr. 2016 Jan-Feb;16(1):48-61. doi: 10.5698/1535-7597-16.1.48. PMID 26900382
- [Background] McKenzie KC, Hahn CD, Friedman JN. Emergency management of the paediatric patient with convulsive status epilepticus. Paediatr Child Health. 2021 Jan 21;26(1):50-66. doi: 10.1093/pch/pxaa127. eCollection 2021 Feb. PMID 33552322
- [Background] Singh A, Stredny CM, Loddenkemper T. Pharmacotherapy for Pediatric Convulsive Status Epilepticus. CNS Drugs. 2020 Jan;34(1):47-63. doi: 10.1007/s40263-019-00690-8. PMID 31879852
- [Background] Hamano SI, Sugai K, Miki M, Tabata T, Fukuyama T, Osawa M. Efficacy, safety, and pharmacokinetics of intravenous midazolam in Japanese children with status epilepticus. J Neurol Sci. 2019 Jan 15;396:150-158. doi: 10.1016/j.jns.2018.09.035. Epub 2018 Oct 4. PMID 30472551
- [Background] Navarro V, Dagron C, Elie C, Lamhaut L, Demeret S, Urien S, An K, Bolgert F, Treluyer JM, Baulac M, Carli P; SAMUKeppra investigators. Prehospital treatment with levetiracetam plus clonazepam or placebo plus clonazepam in status epilepticus (SAMUKeppra): a randomised, double-blind, phase 3 trial. Lancet Neurol. 2016 Jan;15(1):47-55. doi: 10.1016/S1474-4422(15)00296-3. Epub 2015 Nov 28. PMID 26627366
- [Background] Alvarez V, Rossetti AO. Monotherapy or Polytherapy for First-Line Treatment of SE? J Clin Neurophysiol. 2016 Feb;33(1):14-7. doi: 10.1097/WNP.0000000000000217. PMID 26840871
- [Background] Lynch BA, Lambeng N, Nocka K, Kensel-Hammes P, Bajjalieh SM, Matagne A, Fuks B. The synaptic vesicle protein SV2A is the binding site for the antiepileptic drug levetiracetam. Proc Natl Acad Sci U S A. 2004 Jun 29;101(26):9861-6. doi: 10.1073/pnas.0308208101. Epub 2004 Jun 21. PMID 15210974
- [Background] Klitgaard H, Pitkanen A. Antiepileptogenesis, neuroprotection, and disease modification in the treatment of epilepsy: focus on levetiracetam. Epileptic Disord. 2003 May;5 Suppl 1:S9-16. PMID 12915336
- [Background] Misra UK, Kalita J, Maurya PK. Levetiracetam versus lorazepam in status epilepticus: a randomized, open labeled pilot study. J Neurol. 2012 Apr;259(4):645-8. doi: 10.1007/s00415-011-6227-2. Epub 2011 Sep 6. PMID 21898137
- [Background] Sharpe C, Reiner GE, Davis SL, Nespeca M, Gold JJ, Rasmussen M, Kuperman R, Harbert MJ, Michelson D, Joe P, Wang S, Rismanchi N, Le NM, Mower A, Kim J, Battin MR, Lane B, Honold J, Knodel E, Arnell K, Bridge R, Lee L, Ernstrom K, Raman R, Haas RH; NEOLEV2 INVESTIGATORS. Levetiracetam Versus Phenobarbital for Neonatal Seizures: A Randomized Controlled Trial. Pediatrics. 2020 Jun;145(6):e20193182. doi: 10.1542/peds.2019-3182. Epub 2020 May 8. PMID 32385134